CLINICAL TRIAL: NCT06080659
Title: Network-based biOmarker Discovery of Neurodegenerative Diseases Using Multimodal Connectivity
Acronym: NODAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC22_9712_NODAL
Record Dates: First submitted 2023-09-22; First posted 2023-10-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease, Early Onset; Parkinson Disease
Keywords: connectome
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- DCS+ (Experimental): Patient with subjective cognitive decline, prodromal condition of Alzheimer's disease
  Interventions: Diagnostic Test: fMRI; Diagnostic Test: CONFMEM
- TCL-MA (Experimental): Patient with mild neurocognitive disorder linked to Alzheimer's disease
  Interventions: Diagnostic Test: fMRI; Diagnostic Test: CONFMEM
- MPdn (Experimental): early-stage or de novo Parkinson's disease patients with no cognitive deficits
  Interventions: Diagnostic Test: fMRI; Diagnostic Test: CONFMEM
- TCL-MP (Experimental): Patient with mild neurocognitive disorder linked to Parkinson's disease
  Interventions: Diagnostic Test: fMRI; Diagnostic Test: CONFMEM
- Healthy volunteers (Active Comparator): Healthy volunteers
  Interventions: Diagnostic Test: fMRI; Diagnostic Test: CONFMEM

INTERVENTIONS:
Diagnostic Test: fMRI — functional MRI
Diagnostic Test: CONFMEM — The aim of this paradigm is to identify the impact of cognitive conflict situations on recognition memory (the ability to judge whether or not a stimulus has been previously presented).

SUMMARY:
The aim of the NODAL clinical trial is to demonstrate the feasibility of new, low-cost, non-invasive biomarkers of neurodegenerative pathologies as early Alzheimer and Parkinson, based on the estimation of the multimodal connectome.

DETAILED DESCRIPTION:
Alzheimer's (AD) and Parkinson's (PD) diseases are characterized by pre-clinical and asymptomatic phases, which can extend over decades, before progressing through different clinical stages where cognitive and/or motor symptoms appear. A major challenge for clinical neuroscience is the availability of reliable, non-invasive and inexpensive biomarkers to enable early diagnosis, be clinically relevant, and ideally contribute to prognosis and patient monitoring.

Current criteria, which are essentially clinical, have a relatively low diagnostic accuracy, which is unfortunately responsible for a delay in diagnosis, whereas it has been established that early diagnosis makes it possible to postpone the loss of autonomy, open up opportunities for clinical trials for patients, and, epidemiologically speaking, ultimately reduce the prevalence of major neurocognitive disorders.

Recent advances in neuroimaging techniques and connectome analysis have led to the identification of innovative biomarkers that reflect the disorganization of brain networks and are associated with clinical symptoms.

After participant inclusion, the experimental visit will take place over half a day, for patients with early-stage Alzheimer's or Parkinson's disease and for healthy control volunteers.

After clinical assessment, participants will undergo an MRI scan and then perform the CONFMEM experimental task.

The aim of this paradigm is to identify the impact of cognitive conflict situations on recognition memory (the ability to judge whether or not a stimulus has been previously presented).

The cerebral connectome will be assessed for each patient, with the aim of determining whether patterns can lead to pathology-specific markers.

ELIGIBILITY:
Inclusion Criteria:

* For all participants:
* French mother tongue
* right-handed
* with a level of education equal to or higher than the Certificat d'Études Primaires (Primary School Certificate)
* Free of any medical or psychiatric condition likely to interfere with cognition (excluding diagnosis for patients)
* Affiliated with a social security scheme
* Having received oral and written information about the protocol and having signed a consent form to participate in this research.

DCS+ group:

- Meeting the diagnostic criteria for "subjective cognitive decline-plus" (Jessen criteria (Jessen et al., 2014).

Alzheimer's patients "Mild Cognitive Impairment due to Alzheimer's Disease," "MCI-MA":

- Meeting the diagnostic criteria for "Mild neurocognitive disorder due to Alzheimer's disease" (criteria of (Albert et al., 2011))

De novo" Parkinsonian patients, "MPdn":

- Presenting with newly diagnosed ("de novo") Parkinson's disease and free of cognitive deficits (criteria of Postuma et al., 2015 (Postuma et al., 2015))

Parkinsonian patients with "Mild Cognitive Impairment, "MCI-MP":

- Presenting Parkinson's disease associated with "mild neurocognitive impairment" (criteria of Litvan et al., 2012 (Litvan et al., 2012))

Exclusion Criteria:

* All participants (healthy volunteers and patients)
* Contraindications to MRI :
* Abdominal circumference + upper limbs sticking to the body > 200 cm;
* Implantable pacemaker or defibrillator;
* Neurosurgical clips;
* Cochlear implants ;
* Neural or peripheral stimulator;
* Intra-orbital or encephalic metallic foreign bodies;
* Endoprostheses fitted less than 4 weeks ago and osteosynthesis devices fitted less than 6 weeks ago;
* Claustrophobia.
* Pregnant or breast-feeding women;
* Adults under legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.

Patients only

* Score >2 on the modified Hachinski scale (Hachinski et al., 2012)
* Dementia according to McKhann criteria (McKhann et al., 2011)
* Sensory deficit interfering with experimental tests

Healthy volunteers only

- Cognitive impairment (MoCA score < 26)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Multimodal connectivity graph metrics across diseases | 2 hours and 30 minutes
  Multi-layer graph combining the functional and structural connectivity will provide an ideal framework for identifying multimodal features. The first layer corresponds to the functional connectivity where links represent the similarity between the fMRI signal from different cerebral regions (i.e. the nodes), using the cross-correlation. The second layer represents the structural connectivity where the edges are the fiber density between the nodes. Topological metrics of graph: 1/ the nodal centrality which quantifies how important a node is within a network, 2/ the betweenness defined as the ratio of the number of the shortest paths comprising the node to the total number of shortest paths in the graph, measures the hub property of the node and 3/ local efficiency which quantify the ability of a network to transmit information at the global and local level, will be compared between patients at-risk for Alzheimer's Disease, patients with Parkinson's Disease and healthy controls.

SECONDARY OUTCOMES:
Multimodal connectivity graph metrics across stages of disease | 2 hours and 30 minutes
  Multi-layer graph combining the functional and structural connectivity will provide an ideal framework for identifying multimodal features. The first layer corresponds to the functional connectivity where links represent the correlation between the fMRI signal. The second layer represents the structural connectivity where the edges are the fiber density between the nodes. Topological metrics of graph: 1/ the nodal centrality which quantifies how important a node is within a network, 2/ the betweenness defined as the ratio of the number of the shortest paths comprising the node to the total number and 3/ local efficiency which quantify the ability of a network to transmit information, will be compared between patients at-risk for Alzheimer's Disease at the Subjective Cognitive Decline stage and at the Mild Cognitive Impairment stage. Similarly, patients with Parkinson's Disease without cognitive impairment and with Parkinson's Disease with Mild Cognitive will be compared.
Correlation between multimodal connectivity graph metrics and cognitive scores | Up to 6 months (maximum delay between the study visit and the collection of standard tasks).
  Cognitive scores will include standard tasks (MOCA, Symbol Digit Modality Test - oral, Digit span, 16-items Free & Cued Selective Reminding Test, 10/36 spatial recall test, Oral Letter-Number Sequencing test, D-KEFS Color-Word Interference Test, Benton Judgment of Line Orientation, CLOX clock-drawing test, Boston Naming Test, Animal fluency) and an experimental recognition memory task. As for the latter, the scores used will be the congruency effect during study (RT in milliseconds), global recognition accuracy, and the effect of congruency on subsequent memory (difference in recognition accuracy between congruent and incongruent trials at study).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves JONIN, PhD, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France